CLINICAL TRIAL: NCT04420741
Title: Efficacy and Safety of 72-hour Infusion of Prostacyclin (1 Nanogram(ng)/ Kilo(kg)/Minute(Min)) in Patients With COVID-19 Induced Pulmonary Endotheliopathy
Brief Title: Infusion of Prostacyclin (Iloprost) vs Placebo for 72-hours in COVID-19 Patients With Respiratory Failure
Acronym: COMBAT-COVID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pär Johansson (Other)
Responsible Party: Sponsor-Investigator, Pär Johansson, Sponsor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COMBAT-COVID-19; 2020-001296-33 (EudraCT Number)
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: COVID-19; Respiratory Failure
Keywords: COVID-19; SHINE; Endotheliopathy
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency | interventions — Iloprost; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomization active/placebo (1:1) parallel arms
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The preparation will be done by an unblinded study nurse at the respective ICU´s, who will be responsible for preparing the investigational drug so that it can be administered in blinded fashion. Iloprost is a colorless fluid that is to be diluted in 0.9% saline. The infusion pump containing diluted active drug and placebo will be identical on how the fluid looks and behaves.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iloprost (Experimental): Patients randomized to active treatment (n=40 patients) will receive continuous infusion of iloprost for 72 hours after inclusion or until discharge to ward or death, whichever comes first.
  Interventions: Drug: Iloprost
- Isotonic saline (Placebo Comparator): Patients randomized to placebo treatment (n=40 patients) will receive continuous infusion of placebo for 72 hours after inclusion or until discharge to ward or death, whichever comes first.
  Interventions: Drug: Isotonic saline

INTERVENTIONS:
Drug: Iloprost — Continuously infusion for 72 hours at 3 ml/hours. Treatment dose 1 ng/kg/min
  Other Names: Ilomedin
  Arms: Iloprost
Drug: Isotonic saline — Continuously infusion for 72 hours at 3 ml/hours
  Arms: Isotonic saline

SUMMARY:
The purpose of this trial is to investigate the efficacy and safety of continuous intravenous administration of low dose iloprost versus placebo for 72-hours, in 80 patients with COVID-19 suffering from respiratory failure. The study hypothesis is that iloprost may be beneficial as an endothelial rescue treatment as it is anticipated to deactivate the endothelium and restore vascular integrity in COVID-19 patients suffering from respiratory failure caused by endothelial breakdown, ultimately improving survival. Given that the pulmonary system, apart from the brain, is the most highly vascularized vital organ in the body, extensive endothelial damage is a central feature of acute respiratory distress syndrome (ARDS) with respiratory failure being the rationale for the current study COMBAT-COVID-19.

DETAILED DESCRIPTION:
Patients with the most severe type of sepsis, those with septic shock have a mortality rate between 30% to 45% due to multiple organ failure. The poor outcome of shocked patients, and especially those with sepsis, may by related to microvascular endothelial dysfunction.

Coronavirus disease 2019 (COVID-19) is an infectious disease caused by coronavirus 2 (SARS-CoV-2) and, thus, being a novel cause of sepsis. The disease was first identified in 2019 in Wuhan, the capital of Hubei, China, and has since spread globally, resulting in the 2019-20 coronavirus pandemic. Common symptoms include fever, cough and shortness of breath, muscle pain and sputum production. While many cases result in mild symptoms, some progress to pneumonia and multi-organ failure. In particular COVID-19 is associated with ARDS with respiratory failure and high mortality.

Evidence support that iloprost infusion significantly improved endothelial function and integrity, The main objective in this trial is to investigate whether continuous infusion of lov dose iloprost at a dose of 1 ng/kg/min for 72-hours is safe and significantly reduce the need of respiratory support in the intensive care unit (ICU) compared to infusion of placebo in patients with COVID-19 induced pulmonary endotheliopathy (SHINE).

Patients that are eligible for this trial will be temporarily incompetent due to acute severe illness relating to respiratory failure, therefore informed consent will be obtained from a scientific guardian. Next-of kin and subsequently the patient will co-sign as soon as possible hereafter. During the trial, patient will be given continuous infusion of low dose iloprost or placebo for 72 hours and additional blood samples will be obtained at baseline and at 24 hours. Follow up on respiratory failure and mortality will be performed on dag 28 and 90.

This trial is conducted in accordance with the Helsinki 2 Declaration and International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use, Guideline for Good Clinical Practice (ICH-GCP) and in compliance with the protocol. As part of the quality assurance on-site monitoring visit will be performed by the an independent GCP-unit including source data verification. Standard Operation Procedure (SOP) to address protocol specific procedures such as data collection and adverse event reporting are developed.

The number of patients participating is based on a power calculation using the data on days alive and free from mechanical ventilation in the ICU within 28 days from a randomized, double blind, placebo controlled clinical trial in patients with acute respiratory distress syndrome ARDS (NTC 02622724).

The number of patients may be increased if required for regulatory approval for this indication.

ELIGIBILITY:
Inclusion Criteria:

* Adult intensive care patients (aged 18 years or above)
* Confirmed COVID-19 infection
* Need for mechanical ventilation (< 72 hours at time of screening)
* Soluble thrombomodulin (sTM) ≥ 4 ng/mL

Exclusion Criteria:

* Withdrawal from active therapy
* Pregnancy (non-pregnancy confirmed by patient being postmenopausal (age 60 or above) or having a negative urine- or plasma-hCG)
* Known hypersensitivity to iloprost or to any of the other ingredients.
* Previously included in this trial or a prostacyclin trial within 30 days
* Consent cannot be obtained
* Life-threatening bleeding defined by the treating physician
* Known severe heart failure (NYHA class IV)
* Suspected acute coronary syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-04-23 (Actual)

PRIMARY OUTCOMES:
Mechanical ventilation free days | Until ICU discharge, maximun 28 days after randomization
  Days alive without mechanical ventilation in the ICU within 28 days

SECONDARY OUTCOMES:
28 and 90-day mortality | Day 28 and 90 after randomization
  Vital status of the patient at day 28 and day 90
Modified Sequential Organ Failure Assessment (SOFA) | Until ICU discharge, maximun 90 days after randomization
  Mean daily modified SOFA score in the intensive care unit (scores for each of five systems range from 0 to 4, with higher scores indicating more severe dysfunction; range score 0-20).
Vasopressor free days | Until ICU discharge, maximun 90 days after randomization
  Days alive without vasopressor in the ICU within 28-and 90 days
Renal replacement free days | Until ICU discharge, maximun 90 days after randomization
  Days without renal replacement in the ICU within 28 -and 90 days
Mechanical ventilation free days | Until ICU discharge, maximun 90 days after randomization
  Days alive without mechanical ventilation in the ICU within 90 days
Serious adverse reactions (SARs) | Until day 7 after randomization
  Numbers of serious adverse reactions within the first 7 days
Serious adverse events (SAEs) | Until day 7 after randomization
  Numbers of serious adverse events within the first 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Anders Perner, MD, PhD, Principal Investigator — Copenhagen University Hospital, Intensive care Unit 4131; Pär I Johansson, MD, DMSc, Study Director — Copenhagen University Hospital, Capital Blood Bank 2034
Locations (5):
- Denmark (5):
  - Dept. of Anaesthesia and Intensive Care, Bispebjerg Hospital, Copenhagen
  - Dept. of Intensive Care, Copenhagen University Hospital, Rigshospitalet, Copenhagen
  - Dept. of Intensive Care, Copenhagen University Hospital Herlev, Herlev
  - Dept. of Anaesthesia and Intensive Care, Nordsjaelands Hospital, Hillerød
  - Dept. of Anaesthesia and Intensive Care, Hvidovre Hospital, Hvidovre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johansson PI, Soe-Jensen P, Bestle MH, Clausen NE, Kristiansen KT, Lange T, Stensballe J, Perner A. Prostacyclin in Intubated Patients with COVID-19 and Severe Endotheliopathy: A Multicenter, Randomized Clinical Trial. Am J Respir Crit Care Med. 2022 Feb 1;205(3):324-329. doi: 10.1164/rccm.202108-1855OC. PMID 34813414
- [Result] Johansson PI, Bestle M, Soe-Jensen P, Kristiansen KT, Stensballe J, Clausen NE, Perner A. The effect of prostacyclin (Iloprost) infusion at a dose of 1 ng/kg/min for 72 hours compared to placebo in mechanically ventilated patients with COVID-19: A structured summary of a study protocol for a randomized controlled trial. Trials. 2020 Aug 26;21(1):746. doi: 10.1186/s13063-020-04696-2. PMID 32847626